CLINICAL TRIAL: NCT06540053
Title: The Effect of Active Static Hamstring Stretching Exercises on Lumbar Muscle Activation in Office Workers
Brief Title: The Effect of Hamstring Stretching on Lumbar Muscle Activation in Officers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assoc. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 005-HsR
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Office Workers; Muscle Tightness; Lumbar Region; Muscle Shortness; Stretch; Hamstring Flexibility
Keywords: Muscle Activation; Electromyographic Muscle Activity; Stabilization; Viscoelastic Properties; Hamstring Flexibility; Posture; Low back
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Active Static Hamstring Stretching Participants will perform 10-minute active static hamstring exercises for 5 days a week over a period of 6 weeks.
  Interventions: Other: Active Static Hamstring Stretch Exercise
- Control Group (Other): Participants will receive training on spinal protection principles within the office setting and will be sent short messages containing information on maintaining proper posture throughout the day on their phones for a period of 6 weeks.
  Interventions: Other: Waiting List

INTERVENTIONS:
Other: Active Static Hamstring Stretch Exercise — In the first session, participants will be instructed on the principles of spinal protection. Following this, members of the experimental group will engage in active hamstring exercises within the office environment. These exercises will be conducted for 10 minutes, consisting of 10 repetitions of 30-40 seconds of stretching followed by 30 seconds of rest, five days a week for six weeks. Participants in the experimental group will be remotely supervised during the stretching exercises.
  Arms: Study Group
Other: Waiting List — Participants will receive workplace training on spine protection principles and subsequently be placed on a waiting list. Throughout this process, individuals in the designated group will receive text messages on Mondays, Wednesdays, and Fridays over the course of six weeks. These messages will contain information aimed at assisting them in maintaining correct posture throughout the workday.
  Arms: Control Group

SUMMARY:
Prolonged periods of desk work and static postures in office workers lead to various musculoskeletal issues in both the lower and upper extremities. One such issue is hamstring muscle tightness observed in individuals. Tight hamstring muscles contribute to increased electromyographic muscle activity in the lumbar region, altered lumbopelvic rhythm, and changes in lumbar stabilization, leading to low back pain. The viscoelastic properties of the hamstring muscles play a crucial role in maintaining posture and stabilizing the lumbar region. Insufficient hamstring flexibility or viscoelastic properties can alter pelvic position and result in excessive stress in the lumbar region, thereby increasing the risk of low back pain.

It is anticipated that the activation, stabilization, and viscoelasticity of the muscles in the lumbar region will change through static active hamstring stretching exercises, which aim to restore the length-tension relationship in the hamstring muscles. This study aims to investigate the effect of active static hamstring stretching exercises on lumbar muscle activation, stabilization, and viscoelasticity in office workers.

DETAILED DESCRIPTION:
Most office workers spend long hours working at a computer, leading to prolonged periods of sitting. As a result, low back pain is frequently observed among office workers due to extended sitting durations. Issues arising in the lumbar region significantly reduce individuals' quality of life and are the second leading cause of work absenteeism, thus increasing treatment costs.

The movement of the spine occurs through the coordinated functioning of muscles and nerves. While agonist muscles initiate and maintain movement, antagonist muscles control and modulate it. Healthy spinal movements are ensured by the optimal functioning of these muscles. To achieve this, individuals are provided with ergonomic training, core strengthening exercises, and stretching exercises.

The hamstring muscle contributes to the stabilization of the hip and pelvis joints, thereby aiding in the stabilization of the lumbar spine. The relationship between the viscoelastic properties of the hamstring muscle and the lumbar region encompasses a wide range of issues, including low back pain, postural disorders, and pelvic stability. Studies have reported that a minimum of 5-7 hours of sitting leads to hamstring muscle tightness. Hamstring tightness not only reduces the range of motion but also leads to various musculoskeletal problems. The tightness in the hamstring muscles can affect pelvic mobility and lumbopelvic rhythm. Additionally, research has shown a positive relationship between hamstring tightness and the severity of low back pain. Tight hamstring muscles can increase the tension in the muscles and ligaments of the lumbar region, resulting in significantly higher compression loads on the lumbar spine. Other postural changes associated with hamstring tightness may indirectly affect sacroiliac joint stability. Therefore, the flexibility of the hamstring muscles is extremely important for overall health and optimal physical fitness.

Participants will be divided into two groups: control and experimental. Participants will be randomized, stratified by gender, and a total of 50 individuals are planned to participate in the study. The study will last a total of 6 weeks. At the beginning of the study, both groups will receive briefings. The control group will receive training on spinal protection principles within the office. Additionally, participants in this group will receive short text messages on their phones containing information on maintaining proper posture throughout the day, sent on Mondays, Wednesdays, and Fridays for 6 weeks.

The experimental group, in addition to the spinal protection principles training, will perform active static hamstring stretching exercises in the office environment, consisting of 10 repetitions of 30-40 seconds of stretching and 30 seconds of rest, for a total of 10 minutes per session, 5 days a week. Participants in the experimental group will be supervised during the stretching exercises.

To ensure participants' eligibility according to the inclusion and exclusion criteria, the International Physical Activity Questionnaire-Short Form will be administered. The primary outcome measures of the study are electromyographic muscle activity, stabilization, and viscoelastic properties; the secondary outcome measures are myoton, sit-and-reach test, and photographic posture analysis. Assessments will be conducted on a single day and will be performed twice, at the beginning and at the end of the study, by the same researcher who is blinded to the treatment method.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 20 and 50 years
* Who are office workers
* Spending at least 5 hours daily sitting at a desk
* Willing to participate in the study
* And classified as physically inactive according to the International Physical Activity Short Form

Exclusion Criteria:

* Individuals with a history of lumbar spine and knee surgery within the last 6 months
* A history of any hamstring muscle injury within the last 6 months
* Presence of osteoporosis
* Concurrent mental, metabolic, rheumatologic, neuromuscular, cardiovascular, or pulmonary conditions
* Currently pregnant
* And individuals classified as obese (BMI > 30 kg/m²)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Surface Electromyograph | 6 weeks
  The electromyographic muscle activity of the rectus abdominis, erector spinae, internal and external oblique muscles will be evaluated. Muscle contraction activations will be measured using a two-channel Delsys Trigno Avanti Wireless surface EMG system (Delsys, Inc., Boston, MA, USA). Surface EMG electrodes will be used with the Trigno Avanti EMG sensor, placed at the motor points of the muscles. EMG data sampling will be conducted at a rate of 1000 Hz, with a bandwidth of 20-400 Hz, common mode rejection ratio greater than 80 dB, and root mean square calculated using EMG Works 4.0 analysis software (Delsys, Boston, MA, USA). Prior to electrode placement, skin will be cleaned according to criteria specified by SENIAM for the non-invasive assessment of muscles using Surface Electromyography.
Stabilizer Pressure Biofeedback Unit | 6 weeks
  Participants will be assessed using "The Stabilizer Pressure Biofeedback Unit" (Chattanooga Group, Inc., US). The pressure cell of the device will be positioned under the lumbar vertebrae, aligned with the midpoint of the posterior superior iliac spines (PSIS). After inflating the manometer to 40 mmHg, participants will be instructed to draw their abdominal wall inwardly. Success is defined as maintaining 40 mmHg pressure without any compensation. Participants will then lie prone, with the pressure cell positioned under the lower abdominal region, aligned with the midpoint of the anterior superior iliac spines (ASIS). After setting the manometer's pressure to 70 mmHg, participants will be asked to contract their muscles. A successful test requires a pressure decrease of 6-10 mmHg. A decrease of less than 2 mmHg, no change, or an increase in pressure indicates muscle inadequacy.
Myoton | 6 weeks
  To measure the viscoelastic properties of the rectus abdominis, erector spinae, internal, and external oblique muscles, the MyotonPRO (Muomeetria Ltd., Tallinn, Estonia) will be used. Participants will lie comfortably in a prone position. The device probe (3mm diameter, polycarbonate) will be positioned perpendicular to the skin projection of the muscle being measured. A fixed pre-load of 0.18 N will be applied to compress the superficial tissues of the skin. Beneath the compressed subcutaneous tissues, a fixed mechanical force of 0.4 N will apply rapid impulses (15ms) by the device. These mechanical impulses induce local and elastic deformation in the measured muscle. After this deformation, the muscle responds with natural damped oscillations as it returns to its initial state, and these oscillations are recorded as an acceleration graph by sensitive accelerometers at the other end of the probe, which operate frictionlessly and precisely.

SECONDARY OUTCOMES:
Myoton | 6 weeks
  To measure the tone, stiffness, and elasticity of the hamstring muscle, the MyotonPRO (Muomeetria Ltd., Tallinn, Estonia) will be utilized. Muscle stiffness (N/m) is associated with the maximum acceleration of oscillation and the tissue deformation recorded by the transducer. The Myotonometer can measure the stiffness of tissues up to 2 cm below the epidermis (Liang et al., 2022). Participants will be rested for 5 minutes before measurement, seated with arms relaxed along the body, and measurements will be taken at the thickest point of the relevant muscles. During measurement, the Myotonometer's testing probe will be positioned vertically on the skin surface. The probe will be pushed to the required depth to initiate measurement, and proper depth will be confirmed by the indicator light on the device turning from red to green.
Sit and Reach Test | 6 weeks
  This test is a valid and reliable measure widely used in clinical settings to assess hamstring flexibility in young adult populations (ICC: 0.92). The participant sits on the floor with their back and head against the wall, legs extended out to a testing platform where the soles of their feet are in full contact and knees are fully extended. During the test, the feet are bare and the platform base is 26 cm long. With hands stacked on top of each other, the participant slowly and controlledly leans forward without bending their knees during expiration. At the maximum reach point, they hold the position for 2 seconds. Measurement is taken from the tip of the third finger, subtracting 26 cm if the measurement falls short or adding if it exceeds, noted against the 26 cm baseline. A measurement below 30 cm indicates loss of flexibility in the hamstring muscles. The test is repeated twice, and the highest value recorded.
PostureScreen Mobile® App | 6 weeks
  For this research, a device running iOS 17.1.2 will be used. The application allows evaluation of individuals' standing posture from right and left lateral angles, as well as their seated posture from a lateral perspective. Compared to normal posture, the application numerically reports deviations. Within the application, specific reference points are marked on captured photographs using a touchscreen interface. These reference points are utilized to determine postural deviation values and their severity. During image capture, the application displays a green cursor when the phone is level. A distance of 1.5 meters between the phone and the participant is maintained to ensure consistent and accurate measurements across all evaluations. Postural deviation values, calculated in centimeters or degrees for each variable, are reported through the software.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpözgen, Assoc. Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)